CLINICAL TRIAL: NCT05707611
Title: Acute Effects of Various Aerobic Exercise on Rhinitis Symptoms in Patients With Allergic Rhinitis.
Brief Title: Acute Effects of Various Aerobic Exercise in Allergic Rhinitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 3
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinits; Cytokines; Aerobic exercise; Rhinitis symptoms
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Running; Swimming

STUDY DESIGN:
Intervention Model Description: Fifteen patients with allergic rhinitis aged 18 - 45 years old. The experiment was a crossover design in which each participant was given three types of exercise: running, cycling, and swimming. The participant perform moderate intensity exercise 30 minutes/time. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-and post-exercise. The dependent variables between pre-test and post-test were analyzed by a paired t-test. The dependent variables between groups were analyzed by independent t-test. One way repeated measures ANOVA was used to compare the variables among exercise. Differences were considered to be significant at p < 0.05.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Running (Experimental): Running on treadmill in moderate intensity for 30 minutes
  Interventions: Other: Running
- Cycling (Experimental): Cycling on ergometer in moderate intensity for 30 minutes
  Interventions: Other: Cycling
- Swimming (Experimental): Swimming in moderate in tensity for 30 minutes
  Interventions: Other: Swimming

INTERVENTIONS:
Other: Running — The participant perform running on treadmill at moderate intensity exercise 30 minutes/time. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-and post-exercise.
  Arms: Running
Other: Cycling — The participant perform cycling on cycle ergometer at moderate intensity exercise 30 minutes/time. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-and post-exercise.
  Arms: Cycling
Other: Swimming — The participant perform swimming at moderate intensity exercise 30 minutes/time. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-and post-exercise.
  Arms: Swimming

SUMMARY:
This study was to investigate the comparison among acute effects of various aerobic exercise on symptoms in allergic rhinitis patients.

DETAILED DESCRIPTION:
Fifteen patients with allergic rhinitis aged 18 - 45 years old. The experiment was a crossover design in which each participant was given three types of exercise: running, cycling, and swimming. The participant perform moderate intensity exercise 30 minutes/time. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-and post-exercise. The dependent variables between pre-test and post-test were analyzed by a paired t-test. The dependent variables between groups were analyzed by independent t-test. One way repeated measures ANOVA was used to compare the variables among exercise. Differences were considered to be significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of allergic rhinitis diseases
* Clinical symptoms of persistent rhinitis (nasal congestion, sneeze, nasal itching, and running nose) for more than 4 days per week.
* Positive skin prick test (wheal diameter>3 mm.) to house dust mite (D. pteronyssinus) and using normal saline as the negative control.
* Stopped taking all medicine before the study such as antihistamine for at least 3 days, oral steroid and nasal steroid for at least 2 weeks and luekotriene receptor antagonist for at least a week prior to the study, but the patients could take pseudo ephedrine.

Exclusion Criteria:

* Asthma, Chronic rhino-sinusitis, Hypertension, Cardiovascular diseases
* A smoking habit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Rhinitis symptom scores change | Change after each exercise immediately
  Nasal symptoms were assessed using Total Nasal Symptom Score (TNSS) questionnaire. The subjects were asked to score symptoms of persistent allergic rhinitis before and after yoga training protocol. The total nasal symptom scores were computed as the sum of four individual nasal symptom scores; nasal congestion, itching, sneezing, and rhinorrhea. The scores ranged from 0 to 3 scale (0=none, 1=mild, 2=moderate, 3= severe)
Cytokine in nasal secretion change | Change after each exercise immediately
  Nasal secretions collection was performed bilaterally with filter paper strips (7x30 mm Whatman No.42, Whatman, Clifton, NJ). Three filter paper strips were sequentially placed on each anterior portion of the inferior turbinate for 10 min. This filter paper strips were collected into appropriate tubes and centrifuged at 3,000 rpm for 5 min at 4 °C and immediately frozen at -70 °C until later analysis.The levels of cytokines were determined by using Sandwich ELISA technique

SECONDARY OUTCOMES:
Pulmonary functions change | Change after each exercise immediately
  The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration.
Respiratory muscle strength change | Change after each exercise immediately
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds
Peak nasal inspiratory flow change | Change after each exercise immediately
  The subjects placed a mask, which is turned onto a plastic cylinder through which the air passes during inspiration, over the nose and mouth and inspired forcefully through the nose, with lips tightly closed. Inside the cylinder, there is a diaphragm that moves to the airflow, and the maximum peak flow is registered in a scale range from 30-370 L/min. During the procedure, the subjects placed a mask over the nose and mouth and inspired forcefully through the nose, with lips tightly closed.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Result] Aldred S, Love JA, Tonks LA, Stephens E, Jones DS, Blannin AK. The effect of steady state exercise on circulating human IgE and IgG in young healthy volunteers with known allergy. J Sci Med Sport. 2010 Jan;13(1):16-9. doi: 10.1016/j.jsams.2008.07.001. Epub 2008 Oct 31. PMID 18977173
- [Result] Tongtako W, Klaewsongkram J, Jaronsukwimal N, Buranapraditkun S, Mickleborough TD, Suksom D. The effect of acute exhaustive and moderate intensity exercises on nasal cytokine secretion and clinical symptoms in allergic rhinitis patients. Asian Pac J Allergy Immunol. 2012 Sep;30(3):185-92. PMID 23156847
- [Result] Park J, Park JH, Park J, Choi J, Kim TH. Association between Allergic Rhinitis and Regular Physical Activity in Adults: A Nationwide Cross-Sectional Study. Int J Environ Res Public Health. 2020 Aug 5;17(16):5662. doi: 10.3390/ijerph17165662. PMID 32764473